CLINICAL TRIAL: NCT05079893
Title: Influence of Kinesiophobia on Pain Intensity, Disability, Muscle Endurance and Position Sense in Subjects With Chronic Low Back Pain- A Case Control Study
Brief Title: Influence of Kinesiophobia on the Outcome of Chronic Low Back Pain Condition
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB/COHS/FAC/03/May-2021
Record Dates: First submitted 2021-09-23; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Low Back Pain
Keywords: Low back pain; Kinesiophobia; position sense; Endurance
MeSH Terms: conditions — Low Back Pain; Kinesiophobia | interventions — Case-Control Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: The cases will be the patients suffering from low back pain for at least three months and referred by an orthopedic doctor or general physician.
  Interventions: Other: Case control study
- Controls: The controls will be the patients matched for age, sex, handedness who had no complaints of lower back pain
  Interventions: Other: Case control study

INTERVENTIONS:
Other: Case control study — Observational case control study

SUMMARY:
Though large body of evidence reported association between pain and kinesiophobia, there are paucity of studies in associating kinesiophobia to muscle endurance and position sense in patients with Chronic lower back pain [CLBP]. To the best of Investigator's knowledge, till date there is no studies assessing the relationship between kinesiophobia and endurance and position sense in subjects with CLBP. Therefore, the current study aims to compare the impact of kinesiophobia on lumbar extensor endurance, position sense in patient with CLBP and asymptomatic individuals.

DETAILED DESCRIPTION:
Background:

Patients with chronic low back pain (CLBP) frequently present with kinesiophobia. Recent high quality studies reported a moderate to strong evidence of associations between a greater degree of kinesiophobia and greater levels of pain, greater levels of disability and poorer quality of life. However, there are paucity of studies in associating kinesiophobia to muscle endurance and position sense in patients with CLBP.

Objective:

The primary aim of the study is to compare the impact of kinesiophobia on lumbar extensor endurance, position sense in patient with CLBP and asymptomatic individuals. Secondarily, to examine the association between kinesiophobia and lumbar extensor endurance, position sense, pain intensity and functional ability in patients with CLBP. Thirdly to assess the degree of association with various factors on CLBP, lumbar endurance and position sense.

Material and Methods:

This case-control study will have 200 patients with CLBP and 400 controls. Kinesiophobia will be assessed with Tampa Scale for Kinesiophobia. Lumbar endurance will be assessed with Soren's lumbar extensor test and lumbar position sense with neutral and target lumbar re-positioning tests. Secondarily, the pain intensity will be assessed with visual analog scale, functional ability with patient-specific Functional Scale in patients with CLBP. Kinesiophobia, lumbar endurance, and joint position sense will be compared between patients and controls. Kinesiophobia scores will be correlated with lumbar extensor endurance and proprioception joint position errors, pain intensity, and functional ability. Simple and multiple binary logistic regression will be used to determine crude and adjusted Odd's Ratio for kinesiophobia, lumbar position sense and kinesiophobia, lumbar endurance.

ELIGIBILITY:
Inclusion Criteria for CLBP subjects:

* Adults aged between 18 and 50 years.
* Suffering from low back pain for at least three months and referred by an orthopedic doctor or general physician.
* Enough physical autonomy to participate in the physical activities required by the study.

Exclusion Criteria CLBP subjects:

* Low back pain patients with radiculopathy, post fractures, stenosis and history of tumors, cauda equina syndrome and infection.
* Patient under antidepressive medication Inclusion Criteria for Asymptomatic subjects Age 18 years and above, Either gender.

Exclusion Criteria for Asymptomatic subjects

* H/o previous lower back injury.
* H/o lower limb or trunk pathology.
* Presence of deformity, or condition that may alter motor control.
* History of inflammatory, infectious disease and malignancy in the spine
* Patient under anti depressive medication

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Suffering from low back pain for at least three months and referred by an orthopedic doctor or general physician.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Measuring Kinesiophobia. | 5 MONTHS
  Fear of movement/injury or reinjury will be assessed using the Tampa Scale for Kinesiophobia (TSK), a 17 self-reporting items with scores ranging from 17 (absence of fear) to 68 (highest fear). Tampa Scale for Kinesiophobia has been reported to have good reliability in patients with CLBP.
Measuring Lumbar extensor endurance. | 5 MONTHS
  The subjects will be tested during a 1-hour session and will be asked to undergo a body weight dependent isometric back extension (Sorensen) test on a horizontal table
Measuring Lumbar repositioning tests | 5 MONTHS
  Lumbar repositioning tests will be measured with dual inclinometer

SECONDARY OUTCOMES:
Measuring Pain | 5 MONTHS
  measured with Visual analog scale (VAS). The visual analogue scale consists of a 10-cm line, with the left extremity representing (absence of pain) and the right extremity indicating (great pain). Participants were asked to indicate in the scale their current level of pain, higher values being related to more intense pain.
Measuring Functional ability | 5 MONTHS
  Functional ability will be measured using Patient-specific Functional Scale. Patients are asked to rate (on an 11-point scale) the current level of difficulty associated with each activity, where "0" represents "unable to perform" and "10" represents "able to perform at prior level

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Praveen Kumar Kandakurthi, PhD, Study Chair — College of Health Sciences, Gulf Medical University; Dr. Watson Arulsingh Daniel Ragland, PhD, Principal Investigator — College of Health Sciences, Gulf Medical University; Sharad Patil, MPT, Principal Investigator — Thumbay Physical Therapy and Rehabilitation Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kandakurti PK, de Sa Ferreira A, Calazans Nogueira LA, Arulsingh Daniel Ragland W, Patil SS. Influence of kinesiophobia on lumbar position sense in patients with chronic low back pain-a case-control study. J Back Musculoskelet Rehabil. 2025 Sep;38(5):1158-1164. doi: 10.1177/10538127251326152. Epub 2025 Mar 20. PMID 40111910
- [Derived] Kandakurti PK, Arulsingh W, S Patil S. Influence of kinesiophobia on pain intensity, disability, muscle endurance, and position sense in patients with chronic low back pain-a case-control study. Trials. 2022 Jun 6;23(1):469. doi: 10.1186/s13063-022-06406-6. PMID 35668498
- See also: Related Info — https://docs.google.com/document/d/1-fqZdfqfWEFOnx8vHBBICznoQoOIck-cab7iux0cFGE/edit?usp=sharing